CLINICAL TRIAL: NCT06807775
Title: Effects of Time-Restricted Feeding Pattern (16:8) on Metabolic Variables and Appetite Related Gastrointestinal Hormones in Women With Polycystic Ovary Syndrome
Brief Title: Time Restricted Feeding Model in Women With Polycystic Ovary Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aylin Acikgoz Pinar, Associated Proffessor Doctor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-AKD-28; TSA-2024-21146 (Other Grant/Funding Number: Hacettepe University Scientific Research Projects)
Record Dates: First submitted 2025-01-17; First posted 2025-02-04 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-01

CONDITIONS: Polycystic Ovarian Syndrome (PCOS)
Keywords: Polycystic ovary syndrome; 16:8 time-restricted feeding; metabolic risk factors; appetite regulation; obesity
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PCOS+TRF (Experimental): Women with PCOS following time-restricted feeding model (16:8) for 12 weeks
  Interventions: Other: Dietary Intervention (time-restricted feeding model (16:8))
- PCOS+ER (Experimental): Women with PCOS following energy-restricted diet for 12 weeks
  Interventions: Other: Dietary Intervention (energy restricted dietary intervention)
- Control+TRF (Experimental): Healthy women following time-restricted feeding model (16:8) for 12 weeks
  Interventions: Other: Dietary Intervention (time-restricted feeding model (16:8))

INTERVENTIONS:
Other: Dietary Intervention (time-restricted feeding model (16:8)) — Time-Restricted Feeding (16:8 model): Participants can consume food in any amount during an 8-hour window (08:00-16:00), but no food or energy-containing drinks are allowed during the remaining 16-hour fasting period.
  Other Names: Dietary Intervention (Energy Restricted Diet)
  Arms: Control+TRF; PCOS+TRF
Other: Dietary Intervention (energy restricted dietary intervention) — Participants' daily energy needs are calculated based on their basal metabolic rate and physical activity. The energy intake is then reduced by 15-25%. The diet plan consists of 3 main meals and 2-3 snacks, with the daily intake of carbohydrates, proteins, and fats making up 50-60%, 15-20%, and 25-30% of the total daily energy, respectively.
  Arms: PCOS+ER

SUMMARY:
This study aims to evaluate the effects of a 16:8 time-restricted feeding (TRF) model on anthropometric, metabolic, and hormonal parameters in women with polycystic ovary syndrome (PCOS). In addition, the study will assess participants' food preferences, nutrient intake, and gastrointestinal hormone responses, alongside serum glucose, insulin, and glucagon levels, during ad libitum breakfast meals served at the beginning and end of the intervention.

The study consists of three groups: women with PCOS following a 16:8 TRF model for 12 weeks, women with PCOS following an energy-restricted diet for 12 weeks, and healthy women following a 16:8 TRF model for 12 weeks. Women aged 18-40, with PCOS based on the Rotterdam criteria, will be included in the PCOS groups, while those without PCOS-related symptoms will form the control group. Exclusion criteria include pregnancy, lactation, use of hormonal medications, and the presence of comorbidities such as diabetes or severe liver/kidney dysfunction.

Participants in the TRF groups will consume their daily caloric intake within an 8-hour eating window, fasting for the remaining 16 hours, while the energy-restricted group will follow a balanced diet without timing restrictions. Adherence to the dietary interventions will be monitored through weekly 24-hour dietary records. At baseline, participants will complete a demographic questionnaire, receive nutritional education for their nutritional plan, and undergo assessments for anthropometric and blood pressure measurements, sleep quality, food cravings, and physical activity. Biochemical analyses will evaluate thyroid and sex hormones, electrolytes, liver enzymes, lipid profiles, and hemograms. Additionally, all participants will wear smart wristbands (FitBit Charge 5) throughout the study to track sleep and physical activity.

At the beginning and end of the study, participants will consume a standardized ad libitum breakfast meal during the early follicular phase (days 2-5 of menstrual bleeding). Participants will have 30 minutes to eat as much as they wish, and their consumption will be recorded by a dietitian. The nutrient content of the consumed foods will be analyzed using the Nutrition Information System (BEBIS) software. Blood samples will be collected and visual analogue scala (VAS) will be filled at fasting and at 30, 60, 90, and 120 minutes post-meal. Serum glucose, insulin, glucagon, ghrelin, and incretin hormones will be analyzed using the enzyme-linked immunosorbent analysis (ELISA) method.

Data analysis will be performed using SPSS 23.0 via appropriate statistically analysis. Statistical significance is set at p<0.05.

DETAILED DESCRIPTION:
This study aims to investigate the effects of the 16:8 time-restricted feeding (TRF) model on anthropometric, hormonal, metabolic variables, and dietary habits in women with polycystic ovary syndrome (PCOS). The research will evaluate food cravings, food preferences, energy, and macro-micronutrient intake, as well as postprandial responses of glucose, insulin, glucagon and gastrointestinal hormones involved in appetite regulation (ghrelin, glucagon-like peptide (GLP)-1, and gastric inhibitory peptide (GIP)) in women with PCOS. The findings will be compared to a group of women with PCOS following an energy-restricted diet model and a control group of healthy women adhering to the 16:8 time-restricted feeding model.

The study will include adult women who were newly diagnosed with PCOS according to the Rotterdam criteria (presence of at least two of the following: (I) oligo- or anovulation, (II) clinical or biochemical hyperandrogenism, and (III) polycystic ovary morphology on ultrasound) or who had previously been diagnosed with PCOS but had not undergone any medical or nutritional therapy. Participants will be recruited from the Endocrinology and Metabolism Clinic of Hacettepe University Faculty of Medicine, Department of Internal Medicine. For the control group, volunteers with no chronic diseases will be recruited via posters announcing the study.

The study will include the following groups:

(I) Women with PCOS following time-restricted feeding model (16:8) for 12 weeks (II) Women with PCOS following an energy-restricted diet for 12 weeks (III) Healthy women following time-restricted feeding model (16:8) for 12 weeks Due to the lack of similar studies in the literature, an initial sample size of 15 participants per group will be recruited. Interim analysis will be conducted once 15 participants per group are reached. It is expected that participants will lose 5% of their initial body weight after the 12-week dietary intervention, and the interim analysis will be evaluated based on this parameter. If the achieved statistical power is 80% or higher, the study will be concluded; however, if it falls below 80%, the number of additional participants required to reach 80% power will be determined.

For PCOS groups, women aged 19-35 years with body mass index (BMI) 25-40 kg/m2 who meet the diagnostic criteria for PCOS based on the Rotterdam criteria, will be eligible for participation. Further, participants between the ages of 19-35 with BMI 25-40 kg/m2 who do not meet any PCOS diagnostic criteria after endocrinological and gynecological examinations will be included as the control group. For both PCOS groups and control groups, pregnancy, lactation, presence of chronic diseases such as hypertension, diabetes mellitus, cardiovascular diseases, etc., use of hormonal medications, or the presence of comorbidities such as type 2 diabetes mellitus or severe liver/kidney dysfunction will excluded.

Baseline Data Collection Methods:

Participants who meet the eligibility criteria will be included in the study during the early follicular phase (2nd-5th day of menstrual cycles). At baseline, participants will complete a questionnaire assessing general and demographic characteristics. Participants will be randomly assigned in equal numbers to experimental groups.

Before the intervention, anthropometric and blood pressure measurements will be collected. Height and body weight will be measured to calculate BMI. Body weight will be measured using a digital scale (TANITA BC 418) with 0.1 kg sensitivity while participants are in a fasting state and wearing light clothing. Height will be measured without shoes, with participants standing in the Frankfurt horizontal plane. Waist and hip circumferences will be measured using a non-stretchable tape at the midpoint between the lowest rib and iliac crest (for waist circumference) and at the widest part of the hips (for hip circumference). Waist-to-hip ratio and BMI will be categorized based on WHO criteria. Body composition will be assessed using a bioelectrical impedance analyzer (TANITA BC 418).

Blood pressure (systolic and diastolic) will be measured twice using a digital blood pressure monitor after participants rest for 15 minutes in a seated position. The average of the two readings will be recorded.

To calculate participants' energy requirements, physical activity levels will be assessed using the International Physical Activity Questionnaire-Short Form (IPAQ-S). This questionnaire will be administered at baseline (week 0) and at weeks 2, 4, 6, 8, 10, and 12 of the intervention.

Participants' sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI). Food craving levels will be assessed using the Food Craving Questionnaire. This 6-point Likert-type scale consists of nine subscales, with higher scores indicating increased food cravings. The questionnaires will be administered at baseline (week 0) and at weeks 2, 4, 6, 8, 10, and 12.

A semi-quantitative food frequency questionnaire covering the last three months will be administered at baseline. Dietary intake will be analyzed using the "Food and Nutrient Photo Catalog". Daily consumption amounts will be calculated and entered into the Nutrition Information System (BEBIS) software to determine energy, macronutrient, and micronutrient intakes.

Open Buffet Breakfast Meal and Data Collection During This Process (Beginning of the Study) At the beginning of the study, participants will be served ad libitum breakfast meal including boiled eggs, full-fat white cheese, Kashar cheese, cream cheese, salami, sausages, sujuk, white bread, whole wheat bread, simit (Turkish sesame bagel), plain pastry (acma), cheese-filled pastry (pogaca), plain cornflakes, chocolate-flavored cornflakes, tomatoes, cucumbers, red peppers, green peppers, parsley, iceberg lettuce, raisins, dried apricots, sugar, strawberry, sour cherry, and apricot jams, honey, grape molasses, grape molasses-tahini mixture, black olives, green olives, butter, walnuts, raw hazelnuts, black tea, full-fat cow's milk, orange juice, and mixed fruit juice. The breakfast will be provided to participants during the early follicular phase (between days 2 and 5 of menstrual bleeding). Participants will be informed that they may consume as much as they desire from the available food items, with the breakfast duration limited to 30 minutes. While participants consume the meal, a researcher dietitian will record their food consumption. The consumed foods, along with their quantities, will be entered into the Nutrition Information System (BEBIS) program to determine energy, macronutrient, and micronutrient intakes.

Before participants begin consuming the breakfast (at 0 minutes) and at 30, 60, 90, and 120 minutes after the meal, 5 ml of blood samples will be collected. Serum glucose, insulin, glucagon, ghrelin, GLP-1, and GIP levels will be analyzed using Enzyme-Linked Immunosorbent Assay (ELISA) methods. The area under the curve (AUC) will be calculated for glucose, insulin, glucagon, ghrelin, GLP-1, and GIP levels. Additionally, a Visual Analogue Scale (VAS) with four questions will be applied to participants at the time of blood collection (0, 30, 60, 90, and 120 minutes). The VAS allows participants to rate their hunger, satiety, food cravings, and the amount of food they feel they can consume.

Starting the Dietary Intervention Participants will follow the different dietary programs for 12 weeks. In the time-restricted feeding group, participants will be allowed to consume food in any amount for 8 hours between 08:00-16:00, while no food or drinks with energy content can be consumed during the remaining 16-hour fasting period. For the group applying an energy-restricted diet, participants' daily energy requirements will be calculated using basal metabolic rate and physical activity data, and this requirement will be reduced by 15-25% to create a diet plan. The daily intake of carbohydrates, proteins, and fats will be planned to make up 50-60%, 15-20%, and 25-30% of the total daily energy, respectively. The diet plan will consist of 3 main meals and 2-3 snacks, in line with healthy eating recommendations.

Monitoring Participants During the Diet Intervention and Evaluating Adherence Throughout the 12-week intervention, participants will be interviewed at the end of each week, and food intake will be collected through 24-hour food consumption records. The consumed foods, along with their quantities, will be entered into the BEBIS program to determine energy, macro, and micronutrient intake.

Participants will have face-to-face interviews every two weeks (during the 2nd, 4th, 6th, 8th, 10th, and 12th weeks), during which anthropometric measurements and blood pressure measurements will be taken. Furthermore, the Pittsburgh Sleep Quality Index, International Physical Activity Scale-Short Form, and Food Craving Questionnaire will be applied during the 2nd, 4th, 6th, 8th, 10th, and 12th weeks.

End of the Diet Intervention At the end of the 12th week, anthropometric measurements, blood pressure measurements, and 24-hour food consumption records will be collected, and the International Physical Activity Scale, Pittsburgh Sleep Quality Index, and Food Craving Questionnaire will be applied.

Biochemical tests will be evaluated at both the beginning (0th week) and the end (12th week) of the study. Since the routine control interval for women diagnosed with polycystic ovary syndrome (PCOS) is 12 weeks/3 months, biochemical data for these participants will be obtained from patient files. For the healthy control group, biochemical data will be obtained from Hacettepe University Hospitals. The biochemical evaluation will include thyroid hormones profile, sex hormones profile (follicle-stimulating hormone (FSH), luteinizing hormone (LH), estradiol, total testosterone, anti mullerian hormone (AMH), sex hormone binding hormone (SHBG), electrolytes (sodium, potassium, and chlorine), liver enzymes (alanine aminotransferase, aspartate aminotransferase, alkalen phosphatase, and gamma glutamyl transferase), lipid profile (total triglyceride, total cholesterol, low density lipoprotein-cholesterol (LDL-C), very low density lipoprotein-cholesterol (VLDL-C), high density lipoprotein-cholesterol (HDL-C)), hemograms.

Open Buffet Breakfast Meal and Data Collection During This Process (End of the Study) At the end of the 12th week, participants will be served the same breakfast meal as at the beginning of the study. The breakfast will be served to participants during the early follicular phase (between days 2 and 5 of menstrual bleeding). At this point, the food preferences, energy, macro and micronutrient intake, and postprandial responses of gastrointestinal hormones related to appetite will be examined. Similarly, food consumption records during the breakfast and blood samples will be collected, VAS will be filled, as explained in the section on breakfast to be given at the beginning of the study.

Statistical Analysis The data will be analyzed using SPSS 23.0. Normality tests will assess data distribution, presented as mean ± standard deviation or median with range. Differences between independent groups will be tested using t-tests or Mann-Whitney U tests for numerical data and chi-square tests for categorical data. Paired t-tests or Wilcoxon tests will analyze dependent group comparisons. Correlation analyses (Spearman, Pearson, or Eta coefficient) will evaluate relationships. Visual analog scale (VAS) scores and serum levels of glucose, insulin, glucagon, ghrelin, GLP-1, and GIP will be analyzed within the crossover design using repeated measures ANOVA or Friedman test. Statistical significance is set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* For study groups of women diagnosed with polycystic ovary syndrome (PCOS)

  * Aged between 19 and 35 years, with a diagnosis of PCOS
  * No chronic diseases diagnosed by a physician, other than PCOS
  * Body mass index (BMI) between 25 and 40 kg/m²
  * No use of oral contraceptives, insulin sensitizers, or anti-androgen medications in the last three months
* For the healthy control group

  * Aged between 19 and 35 years
  * No diagnosis of chronic diseases
  * Body mass index (BMI) between 25 and 40 kg/m²
  * No use of oral contraceptives, insulin sensitizers, or anti-androgen medications in the last three months

Exclusion Criteria:

* For all study groups:

  * Being in the menopause, pregnancy, or lactation period
  * Having a diagnosis of any chronic disease (e.g., hypertension, diabetes mellitus, cardiovascular disease, etc.) other than PCOS, as determined by a physician
  * Having hyperprolactinemia, congenital adrenal hyperplasia, androgen-secreting tumors, thyroid disorders, Cushing's syndrome, hepatic or renal dysfunction
  * Using antihyperlipidemic, antihypertensive, or glucocorticoid medications
  * Following any specific dietary treatment

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 45 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Changes in body mass index (BMI) | Beginning of the experiment (week 0), 2nd, 4th, 6th, 8th, 10th study weeks and end of the experiment for each participants (week 12).
  BMI will be calculated using weight (kg) and height (m²). Weight and height will be measured separately and used to derive BMI as a single reported outcome.
Changes in serum fasting glucose and lipit profile | Beginning of the experiment (week 0) and end of the experiment for each participants (12th study week)
  Changes in fasting glucose, triglycerides, total cholesterol, low density lipoprotein-cholesterol, and high density lipoprotein-cholesterol (HDL-C) levels will be measured via enzymatic biochemical analysis. All values will be reported in millimolar (mM) and analyzed collectively as metabolic biomarkers.
Changes in appetite-related hormones (insulin, glucagon, ghrelin, glucagon-like peptid-1, and gastric inhibitory peptide) | At both the beginning (week 0) and completion of the experiment for each participant (12th study week) , measurements were taken at the start of the open buffet breakfast and subsequently at the 30th, 60th, 90th, and 120th minutes.
  Changes in insulin, glucagon, ghrelin, glucagon-like peptide-1, and gastric inhibitory peptide levels will be measured via enzyme-linked immunosorbent assay (ELISA kits). All values will be reported in nanomolar (nM) and analyzed collectively as appetite-regulating hormones.

SECONDARY OUTCOMES:
Food craving | Beginning (week 0), week 2, 4, 6, 8, 10, and end of the study (week 12)
  Compare food craving scores (from the Food Craving Questionnaire) at baseline and across the intervention period.
Sleep quality | Beginning (week 0), week 2, 4, 6, 8, 10, and end of the study (week 12)
  Compare sleep quality (from the Pittsburgh Sleep Quality Index) at baseline and across the intervention period.
Physical activity | Beginning (week 0), week 2, 4, 6, 8, 10, and end of the study (week 12)
  Compare physical activity level (from the International Physical Activity Questionnaire - Short Form) at baseline and across the intervention period.
Change in daily energy intake | 0-12 weeks
  Compare changes in daily total energy intake (kcal) at the beginning and end of the intervention.
Blood pressure | Beginning (week 0), week 2, 4, 6, 8, 10, and end of the study (week 12)
  Compare changes in systolic and diastolic blood pressure.
Visual analogue scale score | At both the beginning (week 0) and completion of the experiment for each participant (12th study week) , measurements were taken at the start of the open buffet breakfast and subsequently at the 30th, 60th, 90th, and 120th minutes.
  Compare changes in visual analogue scale score related to hunger, satiety, desire to consume food and the amount of food they can consume.

IPD SHARING:
Plan to Share IPD: Undecided